CLINICAL TRIAL: NCT07355998
Title: Enhancing Communication and Cognitive Resilience in Surgical Trainees Through Medical Improvisation
Brief Title: Medical Improvisation Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 25-44724
Record Dates: First submitted 2026-01-02; First posted 2026-01-21 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Psychosocial Problem

STUDY DESIGN:
Intervention Model Description: A control arm features OHNS residents who continue their standard medical education. The intervention group features OHNS residents who participate in group improvisation training.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Improvisation Group (Experimental): Otolaryngology Residents taking Improvisation Training
  Interventions: Behavioral: Group Online Improvisation Training
- Control Group (Active Comparator): This control group of OHNS residents continues their standard medical education.
  Interventions: Other: Standard Medical Education

INTERVENTIONS:
Behavioral: Group Online Improvisation Training — 3 Online Group Improvisation Training classes led by a professional is offered every other week for 1 hour to the experimental cohort.
  Arms: Improvisation Group
Other: Standard Medical Education — OHNS residents continue the existing standard medical education.
  Arms: Control Group

SUMMARY:
This study offers improvisation training for otolaryngology residents to see if there is any impact on connection, stress, and mood. A control group of otolaryngology residents continues their standard medical education with no improvisation.

ELIGIBILITY:
Inclusion Criteria:

* Otolaryngology Resident at UCSF

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Connection: Social Connectiveness Scale | 6 weeks
  Team dynamics and interpersonal connectedness are assessed using the Social Connectedness Scale. This is a custom survey developed specifically for this study to measure participants' sense of belonging and connection within the residency program. The scale consists of 5 items rated on a 5-point Likert scale. Total scores range from 0 to 25, with higher scores indicating a greater sense of connectedness (better outcome).
Clinical Decision Making Accuracy and Response Time | 6 weeks
  Clinical decision-making under pressure is assessed using the "Intraoperative Vignettes" assessment. This is a computer-based cognitive test comprising 20 Otolaryngology-Head and Neck Surgery (OHNS) case scenarios. Participants are presented with clinical scenarios and must select the correct management decision. The outcome is reported as a composite of accuracy (total number of correct responses) and response time (time taken to select an answer). Accuracy is scored from 0 to 20, with higher scores indicating better clinical decision-making.

SECONDARY OUTCOMES:
Mood (PANAS) | 6 weeks
  Mood is assessed using the Positive and Negative Affect Schedule (PANAS). This is a validated 20-item self-report questionnaire that measures two distinct dimensions of emotion: Positive Affect (10 items) and Negative Affect (10 items). Participants rate items on a 5-point scale ranging from 1 (Very slightly or not at all) to 5 (Extremely). Scores for each subscale range from 10 to 50.
  * Positive Affect: Higher scores represent higher levels of enthusiasm and energy (better outcome).
  * Negative Affect: Higher scores represent higher levels of subjective distress and unpleasurable engagement (worse outcome).
Anxiety and Depression (DASS-21) | 6 weeks
  Psychological distress is measured using the Depression, Anxiety, and Stress Scale-21 (DASS-21). This is a validated 21-item self-report instrument containing three subscales: Depression, Anxiety, and Stress (7 items per subscale). Participants rate how much each statement applied to them over the past week on a 4-point scale ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much or most of the time). Subscale scores are calculated by summing the scores for the relevant items and multiplying by 2.
  * Range: Each subscale ranges from 0 to 42.
  * Interpretation: Higher scores indicate greater severity of symptoms (worse outcome).
Intervention Satisfaction Score (Intervention Arm Only) | 6 weeks
  Participants in the intervention group complete an Intervention Satisfaction Survey to evaluate the curriculum and learner experience. This measure utilizes a Likert scale to assess participant feedback. Items are rated on a 5-point scale from 1 (Not true at all) to 5 (Completely true), with higher scores indicating higher satisfaction (better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Barrett, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No